CLINICAL TRIAL: NCT01288846
Title: Communication About Medication Through the Medication List Coming Into the Hospital With the Patient, Being Changed in the Hospital and Then Returning With the Patient to the Community.
Brief Title: Medication List in and Out of Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Mette Brekke/Professor, University of Oslo
Other Study IDs: MBKF-03-UiO
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-01

CONDITIONS: Febrile Illness; Acute Cardiovascular Disease; Acute Respiratory Disease
Keywords: medication list; changes in medication; prescription medication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acutly ill, Medical ward, consent: group of acutely ill patient who uses three or more drugs, must be able to give consent.

SUMMARY:
30 patients acute hospitalized to medical ward and their medication records are examined. It is to be recorded how the investigators find information about medicine use by the reception when they do not follow the patient. The record of the changes made during hospital stay is examined, whether they are justified in the discharge summaries and whether they are described in the medical list. After a month is to find out if the GP has recorded or possibly rejected changes to medication made in hospital.

DETAILED DESCRIPTION:
Furthermore is to be recorded how the investigators find information about medicine use by the reception when they do not follow the patient and how long it takes to find the right medicine list. The record of the changes made during hospital stay is examined, whether they are justified in the discharge summaries and whether they are described in the medical list. After a month is to find out if the GP has recorded or possibly rejected changes to medication made in hospital.

This shall be recorded in the review of 30 patient with a focus on their medication list and follow them from admission to a month after discharge.

Medicine List in discharge summaries will be compared with medication written in journal during hospital stay and changes described in the text summaries and medication lists should be checked against the same journal.

Medicine list in the municipality one month after discharge shall be compared with discharge summaries and it will be mapped on the GP register, modified and considered if they are valid.

Hypothesis:

Medicine list is missing at admission by > 50% of patients admitted acutely into hospital.

Medicine List at admission, when available, is often incomplete. When the medication list is not available at admission, its content is often incomplete even after the staff at reception have tried to gather information from different sources.

Changes of regular medication is not always present in the discharge summaries. The changes are not always justified in the discharge summaries. The GP often do not correct the medication list in the journal to the discharge summary.

The GP does not give the patient an updated printout of the list at the first medical consultation after admission.

ELIGIBILITY:
Inclusion Criteria:

* acute hospitalized to medical ward
* using three or more drugs, prescription only

Exclusion Criteria:

* not been able to give consent, if too severely ill or not mentally capable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acutely hospitalized patients into medical ward
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Changes in medication | after 2 months
  It is studied when the patient is still in hospital an 1 month after he is at home.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Brekke, professor, Study Director — University of Oslo
Locations (1):
- Sykehuset Innlandet HF Gjøvik, Gjøvik, Norway